CLINICAL TRIAL: NCT04331769
Title: Randomized Clinical Evaluation of the AccuCinch® Ventricular Restoration System in Patients Who Present With Symptomatic Heart Failure With Reduced Ejection Fraction (HFrEF): The CORCINCH-HF Study
Brief Title: Clinical Evaluation of the AccuCinch® Ventricular Restoration System in Patients Who Present With Symptomatic Heart Failure With Reduced Ejection Fraction (HFrEF): The CORCINCH-HF Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5019
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Dilated Cardiomyopathy
Keywords: Heart Failure; Reduced Ejection Fraction; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device group: AccuCinch Ventricular Restoration System (Experimental): Subjects in this arm will receive the AccuCinch Ventricular Restoration System
  Interventions: Device: AccuCinch Ventricular Restoration System
- Control group: Guideline-Directed Medical Therapy (Active Comparator): Subjects in this arm will receive guideline-directed medical therapy (GDMT)
  Interventions: Drug: Guideline-Directed Medical Therapy

INTERVENTIONS:
Device: AccuCinch Ventricular Restoration System — AccuCinch Ventricular Restoration System
  Arms: Device group: AccuCinch Ventricular Restoration System
Drug: Guideline-Directed Medical Therapy — Guideline-Directed Medical Therapy
  Arms: Control group: Guideline-Directed Medical Therapy

SUMMARY:
Prospective, randomized, open-label, international, multi-center clinical study to evaluate the safety and efficacy of the AccuCinch Ventricular Restoration System in patients with heart failure and reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
The CORCINCH-HF Study is a prospective, randomized, open-label, multicenter, international, clinical safety and efficacy investigation of the AccuCinch Ventricular Restoration System.

Subjects will be randomized in a 1:1 ratio:

1. Treatment group: AccuCinch Ventricular Restoration System plus guideline-directed medical therapy (GDMT) (n~200)
2. Control group: Guideline-directed medical therapy (GDMT) (n~200)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-years or older
2. Ejection Fraction: ≥20% and ≤40% measured by transthoracic echocardiography (TTE) and assessed by an echocardiography (echo) core lab
3. LV end-diastolic diameter ≥55 mm measured by TTE and assessed by an echo core lab
4. Symptom Status:

   1. NYHA III,
   2. NYHA ambulatory IV, or
   3. NYHA II with a heart failure hospitalization within the prior 12 months (of signing the consent)
5. Able to complete six-minute walk test with distance between 100 m and 450 m.
6. Diagnosis and treatment for heart failure should be established at least 90 days before the date of consent. Subjects should be on stable, optimally titrated medical therapy for at least 30 days, as recommended according to current guidelines as standard-of-care for Heart Failure therapy, with any intolerance documented.

   1. "Stable" is defined as no more than a 100% increase or a 50% decrease of total daily doses. Medication changes within this range do not require any additional waiting before the screening assessments
   2. When a total daily dose increase or decrease exceeds that which is considered stable, the screening TTE and CT will be postponed 30 days after the medication change
   3. When additional titration is required to optimize a subject's medication that exceeds what is considered stable, the screening TTE and CT will be postponed at least 30 days after achieving the optimal dose (provided the optimal dose remains outside of the stable parameters)
   4. When a dose-for-dose equivalent change in the class of medication change is made, no additional waiting is required before the screening assessments
   5. When a change in class medication change exceeds what is considered stable, OR a new class of medication is added, the screening TTE and CT will be postponed 30 days after the medication change
   6. If an SGLT2 inhibitor is added to a subject's medications, the screening TTE and CT will be postponed at least 30 days after the addition
   7. If an SGLT2 inhibitor dose changes per the stable definition above, no additional waiting is required before the screening assessments
   8. If an SGLT2 inhibitor dose change exceeds what is considered stable, the screening TTE and CT will be postponed at least 30 days after achieving the optimal dose (provided the dose remains outside of the stable parameters)
   9. When applicable, for guideline-directed device-based therapies: a CRT device must be placed > 90 days before the screening TTE and CT, and an ICD must be placed > 30 days before the screening TTE and CT
7. Able and willing to complete all qualifying diagnostic and functional tests, willing to accept blood product transfusion if required and agrees to comply with study follow-up schedule

Exclusion Criteria:

Cardiovascular

1. Myocardial infarction or any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 90 days prior to consent
2. Untreated clinically significant coronary artery disease (CAD) requiring revascularization
3. Fluoroscopic or echocardiographic evidence of severe aortic arch calcification, mobile aortic atheroma, intracardiac mass, thrombus or vegetation
4. Suboptimal ventricular anatomy or wall thickness as determined from screening echocardiography and/or CT scan
5. Heart failure on the basis other than ischemic or non-ischemic dilated cardiomyopathy (e.g., hypertrophic cardiomyopathy, amyloid cardiomyopathy, restrictive cardiomyopathy, uncorrected congenital heart disease, constrictive pericarditis)
6. Hemodynamic instability within 30 days prior to the implant defined as subject requiring inotropic support or mechanical hemodynamic support
7. Any planned cardiac surgery or interventions within the next 180 days post-randomization (including therapeutic right heart procedures)
8. Active bacterial endocarditis
9. Severe RV dysfunction assessed by right heart catheterization (RHC) and/or TTE
10. Fixed pulmonary hypertension with PA systolic pressure >70 mmHg not responsive to vasodilator therapy
11. History of any stroke within the prior 90 days of consent or documented Modified Rankin Scale ≥ 2 disability from any prior stroke

    Valvular
12. Mitral regurgitation grade 3+ (moderate-severe) or 4+ (severe)
13. Untreated degenerative (primary) mitral valve disease (mild prolapse with no need for intervention is allowable)
14. Prior mitral or aortic valve replacement
15. Tricuspid regurgitation grade 4+ (severe)
16. Moderate or severe aortic valve stenosis (AVA less than 1.5 cm2 or peak velocity AV Vmax >300 cm/sec)
17. Aortic regurgitation grade 2+ (moderate), 3+ (moderate-severe), or 4+ (severe)

    Procedural
18. Anatomical pathology or constraints preventing appropriate access/implant of the AccuCinch Ventricular Restoration System (e.g., femoral arteries will not support a 20F Introducer sheath)
19. Renal insufficiency (i.e., eGFR of <25 ml/min/1.73 m2)
20. Subjects in whom anticoagulation during the procedure is contraindicated
21. Subjects in whom 90 days of antiplatelet therapy is contraindicated
22. Known allergy to nitinol, polyester, or polyethylene
23. Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure

    General
24. Life expectancy <1 year due to non-cardiac conditions
25. Currently participating in another interventional investigational study
26. Subjects on high dose steroids or immunosuppressant therapy
27. Female subjects who are pregnant, of child-bearing potential without a documented birth control method, or who are lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-21 (Estimated)

PRIMARY OUTCOMES:
Freedom from device- or femoral artery access-related major adverse events (MAE) | 180 days
  MAE defined as:
  1. All-cause death,
  2. Myocardial infarction,
  3. Stroke,
  4. Need for non-elective cardiovascular surgery,
  5. Worsening of heart-failure requiring mechanical circulatory support for more than 24 hours
  6. Acute kidney injury requiring renal replacement therapy
Change from baseline in Kansas City Cardiomyopathy Questionnaire Quality of Life Questionnaire (KCCQ) Score | 180 days
  Higher scores in the KCCQ reflect better health status
6-Minute Walk Test (6MWT) distance (m) | 180 days
  Change in 6MWT distance (m) from baseline
Freedom from device- or femoral artery access-related major adverse events (MAE) | 365 days
  MAE defined as:
  1. All-cause death,
  2. Myocardial infarction,
  3. Stroke,
  4. Need for non-elective cardiovascular surgery,
  5. Worsening of heart-failure requiring mechanical circulatory support for more than 24 hours
  6. Acute kidney injury requiring renal replacement therapy
A hierarchical composite endpoint of all-cause deaths, left ventricular assist device (LVAD) implants or heart transplants, heart failure hospitalizations, and changes from baseline in Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS) | 365 days
  A hierarchical composite endpoint of number of all-cause deaths, number of left ventricular assist device (LVAD) implants or heart transplants, number of heart failure hospitalizations, and change from baseline in Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS), evaluated using the Win Ratio method

SECONDARY OUTCOMES:
Number of all-cause deaths or all-cause hospitalizations | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
Number of all-cause deaths | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
Number of all-cause hospitalizations | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
Incidence of all serious adverse events, including device- and procedure- related complications | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
Changes from baseline in New York Heart Association (NYHA) functional class | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
Changes from baseline in Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS) | 30 days, 90 days, 365 days, 545 days, 730 days
  Higher scores in the KCCQ reflect better health status
Changes from baseline in 6-Minute Walk Test (6MWT) | 30 days, 90 days, 365 days, 545 days, 730 days
  Measure in meters
Changes in left ventricular ejection fraction (LVEF) from baseline and from post-procedure/pre-hospital discharge as assessed by echo | 30 days, 90 days, 365 days, 730 days
Changes in left ventricular ejection fraction (LVEF) from baseline and from post-procedure/pre-hospital discharge as assessed by echo and CT | 180 days
Changes in left ventricular end-diastolic volume (LVEDV) from baseline and from post-procedure/pre-hospital discharge as assessed by echo | 30 days, 90 days, 365 days, 730 days
Changes in left ventricular end-diastolic volume (LVEDV) from baseline and from post-procedure/pre-hospital discharge as assessed by echo and CT | 180 days
Changes in left ventricular end-systolic volume (LVESV) from baseline and from post-procedure/pre-hospital discharge as assessed by echo | 30 days, 90 days, 365 days, 730 days
Changes in left ventricular end-systolic volume (LVESV) from baseline and from post-procedure/pre-hospital discharge as assessed by echo and CT | 180 days
Rate and number of cardiovascular death events | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
Rate and number of heart failure death events | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
Rate and number of heart failure-related hospitalizations | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days

OTHER OUTCOMES:
Changes from baseline in mitral effective regurgitant orifice area (EROA) | 30 days, 90 days, 180 days, 365 days, 730 days
Changes from baseline in left atrial strain measured by Echo | 30 days, 90 days, 180 days, 365 days, 730 days
Changes from baseline in left ventricular global longitudinal strain measured by Echo | 30 days, 90 days, 180 days, 365 days, 730 days
Changes from baseline in right ventricular free wall longitudinal strain measured by Echo | 30 days, 90 days, 180 days, 365 days, 730 days
Changes from baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) individual domains | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
  Higher scores in the KCCQ reflect better health status
Changes from baseline in EuroQol Five Dimension Five Level (EQ-5D-5L) Quality of Life Questionnaire | 30 days, 90 days, 180 days, 365 days, 545 days, 730 days
  Lower scores in the EQ-5D-5L reflect better health status
Changes from baseline in right ventricular (RV) fractional area change measured by Echo | 30 days, 90 days, 180 days, 365 days, 730 days
  Measured by percent change
Changes from baseline in tricuspid annular plane systolic excursion (TAPSE) measured by Echo | 30 days, 90 days, 180 days, 365 days, 730 days
  Measured in centimeters or millimeters
Changes from baseline in tricuspid regurgitation measured by Echo | 30 days, 90 days, 180 days, 365 days, 730 days
  Measured using effective regurgitant orifice area (mm2) and regurgitant volume (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Study Chair — Columbia University; Ulrich P Jorde, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine; Shmuel Chen, MD, Principal Investigator — New York Presbyterian/Weill Cornell Medicine
Locations (131):
- United States (105):
  - Grandview Medical Group Research, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dignity Health St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Baptist Health Heart Failure & Transplant Institute, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - Scripps Health, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Hartford Health, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - HCA Florida Largo Hospital, Largo, Florida
  - University of Miami, Miami, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Heart Specialists, Louisville, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Ascension Providence Hospital, Southfield, Michigan
  - Metropolitan Heart and Vascular Institute & Mercy Hosp, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - Deborah Heart & Lung, Browns Mills, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - University at Buffalo, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - CUMC/New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Columbia, South Carolina
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - Austin Heart, Austin, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Houston Heart, Houston, Texas
  - Baylor College of Medicine St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UT Health, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Baylor Scott & White, Plano, Texas
  - Methodist Healthcare System, San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - CJW Chippenham Medical Center, Richmond, Virginia
  - Bon Secours St Mary's Hospital, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Valley Health Winchester, Winchester, Virginia
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Republican Scientific and Practical Centre of Cardiology, Minsk, Belarus
- Belgium (2):
  - OLV Heart Centre, Aalst
  - AZ Sint-Jan-Oostende AV Campus Brugge, Bruges
- Czechia (2):
  - St. Anne's University Hospital, Brno
  - Na Homolce Hospital, Prague
- France (3):
  - Hôpital de la Timone, Marseille
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Clinique-Pasteur, Toulouse
- Germany (5):
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg Universitätsklinikum der Medizinischen Hochschule Brandenburg, Bernau
  - Universitätsklinikum Köln (AöR), Cologne
  - CardioVasculäres Centrum, Frankfurt
  - Universitätsklinikum Halle (Saale), Halle
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
- Greece (3):
  - Hygeia Hospital, Athens
  - Onassis Cardiac Surgery Center, Kallithea
  - Interbalkan Medical Hospital of Thessaloniki, Thessaloniki
- Italy (4):
  - A O U Policlinico G. Rodolico - San Marco, Catania, Catania
  - IRCCS Istituto Clinico Humanitas, Milan, Lombardy
  - AOU Città della salute e della Scienza - Ospedale Molinette, Torino, Torino
  - Centro Cardiologico Monzino S.p.a, Milan
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
- Serbia (4):
  - Institute of Cardiovascular Diseases of Vojvodina, Belgrade
  - Institute of Cardiovascular Diseases, Belgrade
  - University Clinical Centre of Serbia, Belgrade
  - University Clinical Center Niš, Niš

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamid N, Jorde UP, Reisman M, Latib A, Lim DS, Joseph SM, Kurlianskaya A, Polonetsky O, Neuzil P, Reddy V, Foerst J, Gada H, Grubb KJ, Silva G, Kereiakes D, Shreenivas S, Pinney S, Davidavicius G, Sorajja P, Boehmer JP, Kleber FX, Perier P, VAN Mieghem NM, Dumonteil N, Leon MB, Burkhoff D. Transcatheter Left Ventricular Restoration in Patients With Heart Failure. J Card Fail. 2023 Jul;29(7):1046-1055. doi: 10.1016/j.cardfail.2023.03.003. Epub 2023 Mar 22. PMID 36958391